CLINICAL TRIAL: NCT01544595
Title: A Multicenter, Double-blind, Randomized Withdrawal Extension Study of Subcutaneous Secukinumab in Prefilled Syringes to Demonstrate Long-term Efficacy, Safety, and Tolerability up to 4 Years in Subjects With Moderate to Severe Chronic Plaque-type Psoriasis Completing Preceding Psoriasis Phase III Studies With Secukinumab
Brief Title: Extension Study of Secukinumab Prefilled Syringes in Subjects With Moderate to Severe Chronic Plaque-type Psoriasis Completing Preceding Psoriasis Phase III Studies With Secukinumab
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAIN457A2302E1; 2012-000533-39
Record Dates: First submitted 2012-02-28; First posted 2012-03-06 (Estimated); Results first posted 2018-12-20 (Actual); Last update posted 2018-12-20 (Actual); Status verified 2018-11

CONDITIONS: Moderate to Severe Plaque-type Psoriasis
Keywords: Psoriasis, inflammatory skin disease; scaly patches; secukinumab (AIN457); Psoriasis Area and Severity Index (PASI); Investigator Global Assessment (IGA) mod 2011
MeSH Terms: conditions — Psoriasis; Dermatitis | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PASI 75 Responders (Placebo Comparator): PASI 75 responders participated in "randomized withdrawal". Subjects who were PASI 75 responders at Week 52 visit of the core studies (e.g.CAIN457A2302 or CAIN457A2303) and have been on secukinumab s.c. 150 mg or 300 mg in core studies were randomized to continue same s.c. doses of secukinumab in PFS or receive placebo every 4 weeks up to Week 152 or until relapse. Participants on first full relapse received loading dose followed by routine dosing with secukinumab s.c. 150 mg or 300 mg regimen.
  Interventions: Drug: Secukinumab (AIN457); Drug: Placebo
- Partial responders (Experimental): Partial responders were not randomized. Subjects who were partial responders at Week 52 visit in core studies (e.g.CAIN457A2302 or CAIN457A2303) and have been on secukinumab s.c. 150 mg or 300 mg in core studies did not participate in the randomized withdrawal. These subjects continued same treatment s.c. dose in PFS (secukinumab s.c. 150 mg or 300 mg) as they were receiving at the time of completing the maintenance period (Week 52) in the core studies.
  Interventions: Drug: Secukinumab (AIN457)

INTERVENTIONS:
Drug: Secukinumab (AIN457) — Secukinumab is a new type of psoriasis medication called a human monoclonal antibody. Monoclonal antibodies are proteins that recognize and bind to unique proteins that your body produces. Secukinumab binds and reduces the activity of a cytokine (a "messenger" protein in the body) called Interleukin 17 (IL-17). IL-17 is believed to be partly responsible for inflammation (pain, swelling, redness). Researchers believe that IL-17 causes symptoms of plaque-type psoriasis like plaques and scales. A product that targets IL-17 therefore may help to relieve these symptoms and conditions.
Drug: Placebo — Placebo
  Arms: PASI 75 Responders

SUMMARY:
This was an extension study of secukinumab prefilled syringes in subjects with moderate to severe chronic plaque-type psoriasis completing preceding psoriasis phase III studies with secukinumab. Subjects on secukinumab at the end of treatment period in phase III studies (e.g., ongoing CAIN457A2302 and CAIN457A2303 and potentially other secukinumab phase III studies) were eligible to join this extension study. This extension study was planned to collect an additional 2 years of long-term efficacy, safety, and tolerability data of secukinumab in either continuous or interrupted therapy (randomized withdrawal period) in subjects showing at least partial response to secukinumab and completing treatment period on secukinumab in previous phase III studies. In this extension study, the prefilled syringe (PFS) liquid formulation of secukinumab were used.

ELIGIBILITY:
Key Inclusion Criteria:

Completed the full study treatment period of 52 weeks in preceding phase III studies, and have been receiving secukinumab treatment during the maintenance phase of the preceding phase III studies, and show at least a partial response (PASI 50 or better) at Week 52 of the preceding phase III studies.

Written informed consent form.

Key Exclusion Criteria:

A protocol deviation in either of the preceding phase III studies which according to the investigator prevented the meaningful analysis of the extension study for the individual subject.

Ongoing use of prohibited psoriasis or non-psoriasis treatments.

Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test (>10 mIU/mL).

Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unwilling to use effective contraception during the study and for 16 weeks after stopping treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1147 (Actual)
Dates: Start 2012-06-19 (Actual); Primary Completion 2017-06-26 (Actual); Study Completion 2017-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (158):
- United States (31):
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Phoenix, Arizona
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Oceanside, California
  - Novartis Investigative Site, Pasadena, California
  - Novartis Investigative Site, San Diego, California
  - Novartis Investigative Site, Colorado Springs, Colorado
  - Novartis Investigative Site, Snellville, Georgia
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, Topeka, Kansas
  - Novartis Investigative Site, Louisville, Kentucky
  - Novartis Investigative Site, Ann Arbor, Michigan
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Rochester, New York
  - Novartis Investigative Site, High Point, North Carolina
  - Novartis Investigative Site, Warren, Ohio
  - Novartis Investigative Site, Oregon City, Oregon
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Duncansville, Pennsylvania
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Novartis Investigative Site, Johnston, Rhode Island
  - Novartis Investigative Site, Charleston, South Carolina
  - Novartis Investigative Site, Kingsport, Tennessee
  - Novartis Investigative Site, Nashville, Tennessee
  - Novartis Investigative Site, Austin, Texas
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, Salt Lake City, Utah
  - Novartis Investigative Site, Norfolk, Virginia
- Argentina (3):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, Mendoza
- Australia (4):
  - Novartis Investigative Site, Kogarah, New South Wales
  - Novartis Investigative Site, Woolloongabba, Queensland
  - Novartis Investigative Site, Carlton, Victoria
  - Novartis Investigative Site, East Melbourne, Victoria
- Belgium (3):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Liège
- Canada (12):
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Surrey, British Columbia
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Moncton, New Brunswick
  - Novartis Investigative Site, Halifax, Nova Scotia
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, Markham, Ontario
  - Novartis Investigative Site, Peterborough, Ontario
  - Novartis Investigative Site, Richmond Hil, Ontario
  - Novartis Investigative Site, Waterloo, Ontario
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Sainte-Foy, Quebec
- Colombia (3):
  - Novartis Investigative Site, Barranquilla, Atlántico
  - Novartis Investigative Site, Barranquilla
  - Novartis Investigative Site, Bogotá
- Estonia (2):
  - Novartis Investigative Site, Tallinn
  - Novartis Investigative Site, Tartu
- Novartis Investigative Site, Helsinki, Finland
- France (7):
  - Novartis Investigative Site, Paris, Cedex 10
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Martigues
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Reims
  - Novartis Investigative Site, Toulouse
- Germany (28):
  - Novartis Investigative Site, Cologne, North Rhine-Westphalia
  - Novartis Investigative Site, Augsburg
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bielefeld
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Darmstadt
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Erfurt
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Gera
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Greifswald
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanau
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Krefeld
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Osnabrück
  - Novartis Investigative Site, Plauen
  - Novartis Investigative Site, Recklinghausen
  - Novartis Investigative Site, Schwerin
  - Novartis Investigative Site, Tübingen
  - Novartis Investigative Site, Wuppertal
- Novartis Investigative Site, Guatemala City, Guatemala
- Hungary (6):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Kaposvár
  - Novartis Investigative Site, Miskolc
  - Novartis Investigative Site, Szeged
  - Novartis Investigative Site, Szombathely
- Novartis Investigative Site, Kopavogur, Iceland
- Israel (3):
  - Novartis Investigative Site, Afula
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Ramat Gan
- Italy (2):
  - Novartis Investigative Site, Catania, CT
  - Novartis Investigative Site, Modena, MO
- Japan (17):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Kurume, Fukuoka
  - Novartis Investigative Site, Maebashi, Gunma
  - Novartis Investigative Site, Asahikawa, Hokkaido
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Kobe, Hyōgo
  - Novartis Investigative Site, Inashiki-gun, Ibaraki
  - Novartis Investigative Site, Isehara, Kanagawa
  - Novartis Investigative Site, Kawasaki, Kanagawa
  - Novartis Investigative Site, Sagamihara, Kanagawa
  - Novartis Investigative Site, Kyoto, Kyoto
  - Novartis Investigative Site, Bunkyo Ku, Tokyo
  - Novartis Investigative Site, Chiyoda-ku, Tokyo
  - Novartis Investigative Site, Minato-ku, Tokyo
  - Novartis Investigative Site, Shinagawa-ku, Tokyo
  - Novartis Investigative Site, Shinjuku-ku, Tokyo
- Latvia (3):
  - Novartis Investigative Site, Daugavpils, LVA
  - Novartis Investigative Site, Ventspils, LVA
  - Novartis Investigative Site, Riga
- Lithuania (3):
  - Novartis Investigative Site, Kaunas, LTU
  - Novartis Investigative Site, Klaipėda, LTU
  - Novartis Investigative Site, Vilnius
- Poland (3):
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Poznan
  - Novartis Investigative Site, Wroclaw
- Novartis Investigative Site, Bucharest, Romania
- Novartis Investigative Site, Singapore, Singapore
- South Korea (6):
  - Novartis Investigative Site, Daejeon, Korea
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul, Seocho-gu
  - Novartis Investigative Site, Busan
  - Novartis Investigative Site, Gwangju
  - Novartis Investigative Site, Seoul
- Spain (5):
  - Novartis Investigative Site, Sabadell, Barcelona
  - Novartis Investigative Site, Santa Coloma de Gramanet, Catalonia
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
- Sweden (2):
  - Novartis Investigative Site, Malmo
  - Novartis Investigative Site, Uppsala
- Taiwan (3):
  - Novartis Investigative Site, Taoyuan District, Taiwan
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taipei
- United Kingdom (7):
  - Novartis Investigative Site, Plymouth, Devon
  - Novartis Investigative Site, London, England
  - Novartis Investigative Site, Salford, Manchester
  - Novartis Investigative Site, Yeovil, Somerset
  - Novartis Investigative Site, Dudley, West Midlands
  - Novartis Investigative Site, Harrogate
  - Novartis Investigative Site, Nuneaton

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Langley RG, Sofen H, Dei-Cas I, Reich K, Sigurgeirsson B, Warren RB, Paul C, Szepietowski JC, Tsai TF, Hampele I, You R, Charef P, Papavassilis C. Secukinumab long-term efficacy and safety in psoriasis through to year 5 of treatment: results of a randomized extension of the phase III ERASURE and FIXTURE trials. Br J Dermatol. 2023 Feb 10;188(2):198-207. doi: 10.1093/bjd/ljac040. PMID 36763857

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Among the 1146 patients who completed the screening phase, 995 "PASI 75 responder at week 52" patients were randomized in a double blind fashion to either active treatment or placebo & entered the randomized withdrawal period and 151 "partial responders at week 52" patients entered treatment period of the Extension.
Pre-assignment Details: 1366 patients who completed the core studies (CAIN457A2302 or CAIN457A2303) and provided consent for participation in the extension study were screened, and 1146 (83.9%) completed the screening phase and entered the extension.
Groups:
- AIN457 150 mg -Randomized Withdrawal Period: PASI 75 responders at Week 52, treated with AIN 150 mg in core study and randomized to AIN150 mg
- AIN457 300 mg -Randomized Withdrawal Period: PASI 75 responders at Week 52, treated with AIN 300 mg in core study and randomized to AIN300 mg
- AIN457 150 mg Placebo - Randomized Withdrawal Period: PASI 75 responders at Week 52, treated with AIN 150 mg in core study and randomized to placebo
- AIN457 300 mg Placebo - Randomized Withdrawal Period: PASI 75 responders at Week 52, treated with AIN 300 mg in core study and randomized to placebo
- AIN457 150 mg - Partial Responders: PASI 50 responders / PASI 75 non responders at Week 52, treated with AIN 150 mg in core and extension study
- AIN457 300 mg - Partial Responders: PASI 50 responders / PASI 75 non responders at Week 52, treated with AIN 300 mg in core and extension study
Period: Status at Week 68
Arm/Group | AIN457 150 mg -Randomized Withdrawal Period | AIN457 300 mg -Randomized Withdrawal Period | AIN457 150 mg Placebo - Randomized Withdrawal Period | AIN457 300 mg Placebo - Randomized Withdrawal Period | AIN457 150 mg - Partial Responders | AIN457 300 mg - Partial Responders
Started | 301 | 363 | 150 | 181 | 0 (These patients were not in the study arms at this time point.) | 0 (These patients were not in the study arms at this time point.)
Completed (Week 68) | 262 | 346 | 87 | 130 | 0 (These patients were not in the study arms at this time point.) | 0 (These patients were not in the study arms at this time point.)
Not Completed | 39 | 17 | 63 | 51 | 0 | 0
Not completed — Adverse Event | 3 | 2 | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Non-compliance with study treatment | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 2 | 0 | 1 | 1 | 0 | 0
Not completed — Technical problems | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 2 | 0 | 0
Not completed — Moved to treatment period ≤ wk 68 | 30 | 13 | 60 | 46 | 0 | 0
Period: Status at Week 156
Arm/Group | AIN457 150 mg -Randomized Withdrawal Period | AIN457 300 mg -Randomized Withdrawal Period | AIN457 150 mg Placebo - Randomized Withdrawal Period | AIN457 300 mg Placebo - Randomized Withdrawal Period | AIN457 150 mg - Partial Responders | AIN457 300 mg - Partial Responders
Started | 301 | 363 | 150 | 181 | 98 | 53
Completed (Week 156) | 184 | 285 | 10 | 15 | 60 | 38
Not Completed | 117 | 78 | 140 | 166 | 38 | 15
Not completed — Withdrawal by Subject | 9 | 10 | 4 | 9 | 20 | 6
Not completed — Adverse Event | 9 | 11 | 1 | 3 | 4 | 2
Not completed — Lost to Follow-up | 4 | 4 | 0 | 1 | 4 | 1
Not completed — Non-compliance with study treatement | 0 | 1 | 0 | 1 | 0 | 1
Not completed — Physician Decision | 0 | 3 | 1 | 0 | 0 | 0
Not completed — Pregnancy | 2 | 3 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 3 | 1 | 2 | 2 | 0 | 0
Not completed — Technical problems | 3 | 1 | 0 | 1 | 0 | 0
Not completed — Moved to treatment period ≤ wk 156 | 86 | 44 | 131 | 145 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 1 | 4 | 10 | 5

BASELINE CHARACTERISTICS:
Population: Randomized set was defined as all patients who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | AIN457 150 mg -Randomized Withdrawal Period | AIN457 300 mg -Randomized Withdrawal Period | AIN457 150 mg Placebo - Randomized Withdrawal Period | AIN457 300 mg Placebo - Randomized Withdrawal Period | AIN457 150 mg - Partial Responders | AIN457 300 mg - Partial Responders | Total
Number analyzed (Participants) | 301 | 363 | 150 | 181 | 98 | 53 | 1146
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.9 (12.93) | 45.8 (12.92) | 47.1 (13.34) | 45.4 (13.09) | 46.8 (12.78) | 48.5 (11.98) | 46.2 (12.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 102 | 45 | 62 | 28 | 10 | 330
  Male | 218 | 261 | 105 | 119 | 70 | 43 | 816
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 213 | 276 | 115 | 136 | 73 | 42 | 855
  Black | 4 | 4 | 2 | 3 | 4 | 1 | 18
  Asian | 52 | 50 | 22 | 24 | 17 | 8 | 173
  Native American | 24 | 23 | 9 | 15 | 2 | 2 | 75
  Pacific Islander | 1 | 2 | 0 | 1 | 1 | 0 | 5
  Unknown | 0 | 1 | 1 | 1 | 0 | 0 | 3
  Other | 7 | 7 | 1 | 1 | 1 | 0 | 17

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants With Loss of Psoriasis Area and Severity Index (PASI) 75 Response up to Week 68
Description: The primary variable was the cumulative rate of patients who lost PASI 75 response up to Week 68 (time=0 being defined as Week 52).
  Loss of PASI 75 response was analyzed by means of a survival analysis defining "loss of PASI 75 response" as "failure". The term cumulative rate corresponded to 1 minus the survival function within this survival analysis, and the cumulative rate and the survival functions were dependent on time t.
  PASI 75 response: patients achieving ≥ 75% improvement (reduction) in PASI score compared to baseline of the core study were defined as PASI 75 responders.
Time Frame: At week 68 (16 weeks after week 52)
Population: Full analysis set (FAS): patients from randomized set with at least 1 post baseline efficacy assessment.
Measure: Number (95% Confidence Interval); unit: Cummulative rate
Arm/Group | AIN457 150 mg -Randomized Withdrawal Period | AIN457 300 mg -Randomized Withdrawal Period | AIN457 150 mg Placebo - Randomized Withdrawal Period | AIN457 300 mg Placebo - Randomized Withdrawal Period
Number analyzed (Participants) | 297 | 363 | 150 | 180
Cummulative rate | 49.8 [25.8 to 79.7] | 25.4 [9.8 to 56.5] | 74.3 [56.9 to 88.8] | 64.7 [52.0 to 77.2]
Statistical Analysis 1: Comparison: AIN457 150 mg -Randomized Withdrawal Period vs AIN457 150 mg Placebo - Randomized Withdrawal Period; The following hypotheses were tested for 52 weeks≤ t ≤68 weeks * H1: p1(t) - p0,1(t) = 0 versus HA1: p1(t)- p0,1(t) ≥ 0, * H2: p2(t) - p0,2(t) = 0 versus HA2: p2(t) - p0,2(t) ≥ 0,; Test type: Superiority — H1: Secukinumab 150 mg was not different from placebo with respect to the cumulative rate for patients who lost PASI 75 response up to Week 68 • H2: Secukinumab 300 mg was not different from placebo with respect to the cumulative rate for patients who lost PASI 75 response up to Week 68; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.30, 95% CI 2-sided [0.22 to 0.42]
Statistical Analysis 2: Comparison: AIN457 300 mg -Randomized Withdrawal Period vs AIN457 300 mg Placebo - Randomized Withdrawal Period; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.20, 95% CI 2-sided [0.14 to 0.29]

2. Secondary Outcome: Number of Participants With PASI 50, PASI 75, PASI 90, PASI 100 and IGA Mod 2011 0 or 1 (Observed Data) - Randomized Withdrawal Period
Description: Psoriasis Area and Severity Index (PASI) 75 responder at week 52. Patients in the placebo groups were not evaluable after re-treatment with Secukinumab.
  PASI 75 Responders: patients with a PASI 75 response (patients achieving ≥75% improvement [reduction] in PASI score compared to baseline of the core study).
  PASI 50 response: patients achieving ≥ 50% improvement (reduction) in PASI score compared to baseline of the core study were defined as PASI 50 responders.
  PASI 90 response: patients achieving ≥ 90% improvement (reduction) in PASI score compared to baseline of the core study were defined as PASI 90 responders.
  PASI 100 response/remission: complete clearing of psoriasis (PASI=0)
Time Frame: Week 52, 104, and 156
Population: FAS
Measure: Number; unit: Number of participants
Arm/Group | AIN457 150 mg -Randomized Withdrawal Period | AIN457 300 mg -Randomized Withdrawal Period | AIN457 150 mg Placebo - Randomized Withdrawal Period | AIN457 300 mg Placebo - Randomized Withdrawal Period
Number analyzed (Participants) | 297 | 363 | 150 | 180
Number of participants
  Wk 52 - IGA 0/1 | 208 | 309 | 112 | 157
  Wk 52 - PASI 50 | 297 | 363 | 149 | 180
  Wk 52 - PASI 75 | 296 | 361 | 149 | 179
  Wk 52 - PASI 90 | 190 | 303 | 105 | 156
  Wk 52 - PASI 100 | 93 | 191 | 54 | 96
  Wk 104 - IGA 0/1: number analyzed (Participants) | 260 | 338 | 20 | 34
  Wk 104 - IGA 0/1 | 128 | 236 | 8 | 13
  Wk 104 - PASI 50: number analyzed (Participants) | 260 | 338 | 20 | 34
  Wk 104 - PASI 50 | 254 | 329 | 19 | 28
  Wk 104 - PASI 75: number analyzed (Participants) | 260 | 338 | 20 | 34
  Wk 104 - PASI 75 | 209 | 299 | 15 | 21
  Wk 104 - PASI 90: number analyzed (Participants) | 260 | 338 | 20 | 34
  Wk 104 - PASI 90 | 125 | 240 | 6 | 13
  Wk 104 - PASI 100: number analyzed (Participants) | 260 | 338 | 20 | 34
  Wk 104 - PASI 100 | 65 | 151 | 4 | 6
  Wk 156 - IGA 0/1: number analyzed (Participants) | 239 | 324 | 10 | 15
  Wk 156 - IGA 0/1 | 90 | 202 | 4 | 7
  Wk 156 - PASI 50: number analyzed (Participants) | 239 | 324 | 10 | 15
  Wk 156 - PASI 50 | 230 | 322 | 10 | 15
  Wk 156 - PASI 75: number analyzed (Participants) | 239 | 324 | 10 | 15
  Wk 156 - PASI 75 | 183 | 287 | 6 | 13
  Wk 156 - PASI 90 (n=239, 324, 10,15): number analyzed (Participants) | 239 | 324 | 10 | 15
  Wk 156 - PASI 90 (n=239, 324, 10,15) | 101 | 207 | 4 | 7
  Wk 156 - PASI 100: number analyzed (Participants) | 239 | 324 | 10 | 15
  Wk 156 - PASI 100 | 47 | 117 | 2 | 5

3. Secondary Outcome: Number of Participants With PASI 50, PASI 75, PASI 90, and PASI 100 (Observed Data) - Entire Study Period
Description: Psoriasis Area and Severity Index (PASI) scoring system: The average degree of severity of each sign in each of the four body regions was assigned a score of 0-4. The area covered by lesions on each body region was estimated as a percentage of the total area of that particular body region.
Time Frame: Week 52, Week 104, Week 156, week 208, week 260
Population: FAS
Measure: Number; unit: Number of participants
Groups:
- AIN457 150 mg Only: patients staying strictly on AIN457 150mg from Week 52
- AIN457 300 mg Only: Patients staying strictly on AIN457 300mg from Week 52
Arm/Group | AIN457 150 mg Only | AIN457 300 mg Only
Number analyzed (Participants) | 164 | 416
Number of participants
  Wk 52 - PASI 50 | 164 | 416
  Wk 52 - PASI 75 | 121 | 361
  Wk 52 - PASI 90 | 85 | 303
  Wk 52 - PASI 100 | 54 | 191
  Wk 104 - PASI 50: number analyzed (Participants) | 104 | 377
  Wk 104 - PASI 50 | 99 | 359
  Wk 104 - PASI 75: number analyzed (Participants) | 104 | 377
  Wk 104 - PASI 75 | 76 | 314
  Wk 104 - PASI 90: number analyzed (Participants) | 104 | 377
  Wk 104 - PASI 90 | 62 | 243
  Wk 104 - PASI 100: number analyzed (Participants) | 104 | 377
  Wk 104 - PASI 100 | 46 | 153
  Wk 156 - PASI 50: number analyzed (Participants) | 69 | 361
  Wk 156 - PASI 50 | 67 | 351
  Wk 156 - PASI: number analyzed (Participants) | 69 | 361
  Wk 156 - PASI | 63 | 297
  Wk 156 - PASI 90: number analyzed (Participants) | 69 | 361
  Wk 156 - PASI 90 | 52 | 211
  Wk 156 - PASI 100: number analyzed (Participants) | 69 | 361
  Wk 156 - PASI 100 | 37 | 118
  Wk 208 - PASI 50: number analyzed (Participants) | 58 | 323
  Wk 208 - PASI 50 | 58 | 316
  Wk 208 - PASI 75: number analyzed (Participants) | 58 | 323
  Wk 208 - PASI 75 | 55 | 269
  Wk 208 - PASI 90: number analyzed (Participants) | 58 | 323
  Wk 208 - PASI 90 | 51 | 194
  Wk 208 - PASI 100: number analyzed (Participants) | 58 | 323
  Wk 208 - PASI 100 | 33 | 104
  Wk 260 - PASI 50: number analyzed (Participants) | 51 | 285
  Wk 260 - PASI 50 | 51 | 279
  Wk 260 - PASI 75: number analyzed (Participants) | 51 | 285
  Wk 260 - PASI 75 | 49 | 231
  Wk 260 - PASI 90: number analyzed (Participants) | 51 | 285
  Wk 260 - PASI 90 | 37 | 179
  Wk 260 - PASI 100: number analyzed (Participants) | 51 | 285
  Wk 260 - PASI 100 | 26 | 100

4. Secondary Outcome: Percent Change From Baseline for PASI Score Over Time (Observed Data) - Randomized Withdrawal Period
Description: The improvement (decrease from baseline) in PASI total scores observed at Week 52.
  Perc. change = 100 x Abs. change /Base. (Abs. change = Post - Base) For each post-baseline visit only patients with a value at both baseline and the respective post-baseline visit are included.
Time Frame: Week 52, 104, and 156
Population: FAS
Measure: Mean (Standard Deviation); unit: Percent change in PASI score
Arm/Group | AIN457 150 mg -Randomized Withdrawal Period | AIN457 300 mg -Randomized Withdrawal Period | AIN457 150 mg Placebo - Randomized Withdrawal Period | AIN457 300 mg Placebo - Randomized Withdrawal Period
Number analyzed (Participants) | 297 | 363 | 150 | 180
Percent change in PASI score
  Week 52 (baseline) | -92.31 (7.878) | -95.98 (6.638) | -92.88 (8.435) | -96.16 (6.030)
  Week 104: number analyzed (Participants) | 260 | 338 | 20 | 34
  Week 104 | -85.88 (14.631) | -91.51 (13.221) | -82.67 (15.568) | -78.04 (20.986)
  Week 156: number analyzed (Participants) | 239 | 324 | 10 | 15
  Week 156 | -83.32 (17.341) | -90.50 (11.660) | -79.77 (15.172) | -86.35 (15.602)

5. Secondary Outcome: Percent Change From Baseline for PASI Score Over Time (Observed Data) - Entire Study Period
Description: Perc. change = 100 x Abs. change /Base. (Abs. change = Post - Base) For each post-baseline visit only patients with a value at both baseline and the respective post-baseline visit are included.
Time Frame: Week 52, Week 104, Week 156, week 208, week 260
Population: FAS
Measure: Mean (Standard Deviation); unit: Percent change in PASI score
Arm/Group | AIN457 150 mg Only | AIN457 300 mg Only
Number analyzed (Participants) | 164 | 416
Percent change in PASI score
  Wk 52 | -85.93 (14.815) | -91.82 (11.889)
  Wk 104: number analyzed (Participants) | 104 | 377
  Wk 104 | -85.97 (18.811) | -88.86 (16.151)
  Wk 156: number analyzed (Participants) | 69 | 361
  Wk 156 | -93.03 (12.338) | -87.78 (15.114)
  Wk 208: number analyzed (Participants) | 58 | 323
  Wk 208 | -95.71 (7.868) | -88.25 (14.496)
  Wk 260: number analyzed (Participants) | 51 | 285
  Wk 260 | -93.65 (9.959) | -88.08 (14.983)

6. Secondary Outcome: Number of Participants in Each IGA Mod 2011 Category (Observed Data)- Randomized Withdrawal Period
Description: Investigator Global Assessment (IGA) mod 2011; scale from 0 - 4. Score 0: Clear (No signs of psoriasis. Post-inflammatory hyperpigmentation could be Present). Score 1: Almost clear (Normal to pink coloration of lesions; no thickening; no to minimal focal scaling), Score 2: Mild (Pink to light red coloration; just detectable to mild thickening; predominantly fine scaling). Score 3: Moderate (Dull bright red, clearly distinguishable erythema; clearly distinguishable to moderate thickening; moderate scaling). Score 4: Severe (Bright to deep dark red coloration; severe thickening with hard edges; severe /coarse scaling covering almost all or all lesions).
  Patients in the placebo groups were not evaluable after re-treatment with Secukinumab
Time Frame: Week 52 (baseline), 104, and 156
Population: FAS
Measure: Number; unit: Number of participants
Arm/Group | AIN457 150 mg -Randomized Withdrawal Period | AIN457 300 mg -Randomized Withdrawal Period | AIN457 150 mg Placebo - Randomized Withdrawal Period | AIN457 300 mg Placebo - Randomized Withdrawal Period
Number analyzed (Participants) | 297 | 363 | 150 | 180
Number of participants
  Wk 52 - clear | 95 | 188 | 56 | 94
  Wk 52 - almost clear | 113 | 121 | 56 | 63
  Wk 52 - mild | 75 | 44 | 33 | 22
  Wk 52 - moderate | 14 | 9 | 4 | 1
  Wk 52 - severe | 0 | 1 | 1 | 0
  Wk 104 - clear: number analyzed (Participants) | 260 | 338 | 20 | 34
  Wk 104 - clear | 66 | 152 | 3 | 4
  Wk 104 - almost clear: number analyzed (Participants) | 260 | 338 | 20 | 34
  Wk 104 - almost clear | 62 | 84 | 5 | 9
  Wk 104 - mild: number analyzed (Participants) | 260 | 338 | 20 | 34
  Wk 104 - mild | 78 | 64 | 9 | 9
  Wk 104 - moderate: number analyzed (Participants) | 260 | 338 | 20 | 34
  Wk 104 - moderate | 47 | 33 | 3 | 10
  Wk 104 - severe: number analyzed (Participants) | 260 | 338 | 20 | 34
  Wk 104 - severe | 7 | 5 | 0 | 2
  Wk 156 - clear: number analyzed (Participants) | 239 | 324 | 10 | 15
  Wk 156 - clear | 48 | 115 | 2 | 4
  Wk 156 - almost clear: number analyzed (Participants) | 239 | 324 | 10 | 15
  Wk 156 - almost clear | 42 | 87 | 2 | 3
  Wk 156 - mild: number analyzed (Participants) | 239 | 324 | 10 | 15
  Wk 156 - mild | 88 | 78 | 2 | 5
  Wk 156 - moderate: number analyzed (Participants) | 239 | 324 | 10 | 15
  Wk 156 - moderate | 59 | 43 | 4 | 2
  Wk 156 - severe: number analyzed (Participants) | 239 | 324 | 10 | 15
  Wk 156 - severe | 2 | 1 | 0 | 1

7. Secondary Outcome: Number of Participants in Each IGA Mod 2011 Category (Observed Data) - Entire Study Period
Description: Investigator's Global Assessment (IGA) mod 2011; scale from 0 - 4. Score 0= clear (no signs of psoriasis) Score 1 = almost clear no to minimal local scaling) Score 2 = mild (predominantly fine scaling) Score 3 = moderate (moderate scaling) Score 4 = severe (severe/coarse scaling covering almost all or all lesions)
Time Frame: Week 52, Week 104, Week 156, week 208, week 260
Population: FAS
Measure: Number; unit: Number of participants
Arm/Group | AIN457 150 mg Only | AIN457 300 mg Only
Number analyzed (Participants) | 164 | 416
Number of participants
  Wk 52 - clear | 56 | 188
  Wk 52 - almost clear | 38 | 123
  Wk 52 - mild | 44 | 71
  Wk 52 - moderate | 26 | 32
  Wk 52 - severe | 0 | 2
  Wk 104 - clear: number analyzed (Participants) | 104 | 377
  Wk 104 - clear | 47 | 154
  Wk 104 - almost clear: number analyzed (Participants) | 104 | 377
  Wk 104 - almost clear | 16 | 85
  Wk 104 - mild: number analyzed (Participants) | 104 | 377
  Wk 104 - mild | 17 | 80
  Wk 104 - moderate: number analyzed (Participants) | 104 | 377
  Wk 104 - moderate | 19 | 51
  Wk 104 - severe: number analyzed (Participants) | 104 | 377
  Wk 104 - severe | 5 | 7
  Wk 156 - clear: number analyzed (Participants) | 69 | 361
  Wk 156 - clear | 37 | 116
  Wk 156 - almost clear: number analyzed (Participants) | 69 | 361
  Wk 156 - almost clear | 13 | 90
  Wk 156 - mild: number analyzed (Participants) | 69 | 361
  Wk 156 - mild | 11 | 91
  Wk 156 - moderate: number analyzed (Participants) | 69 | 361
  Wk 156 - moderate | 8 | 61
  Wk 156 - severe: number analyzed (Participants) | 69 | 361
  Wk 156 - severe | 0 | 3
  Wk 208 - clear: number analyzed (Participants) | 58 | 323
  Wk 208 - clear | 33 | 102
  Wk 208 - almost clear: number analyzed (Participants) | 58 | 323
  Wk 208 - almost clear | 14 | 81
  Wk 208 - mild: number analyzed (Participants) | 58 | 323
  Wk 208 - mild | 7 | 88
  Wk 208 - moderate: number analyzed (Participants) | 58 | 323
  Wk 208 - moderate | 3 | 47
  Wk 208 - severe: number analyzed (Participants) | 58 | 323
  Wk 208 - severe | 1 | 5
  Wk 260 - clear: number analyzed (Participants) | 51 | 285
  Wk 260 - clear | 27 | 97
  Wk 260 - almost clear: number analyzed (Participants) | 51 | 285
  Wk 260 - almost clear | 12 | 65
  Wk 260 - mild: number analyzed (Participants) | 51 | 285
  Wk 260 - mild | 8 | 66
  Wk 260 - moderate: number analyzed (Participants) | 51 | 285
  Wk 260 - moderate | 4 | 53
  Wk 260 - severe: number analyzed (Participants) | 51 | 285
  Wk 260 - severe | 0 | 4

8. Secondary Outcome: Number of Participants With IGA Mod 2011 0/1 Response (Observed Data) - Entire Study Period
Description: Investigator's Global Assessment (IGA) mod 2011 0/1. Score 0= clear (no signs of psoriasis) Score 1 = almost clear no to minimal local scaling) Score 2 = mild (predominantly fine scaling) Score 3 = moderate (moderate scaling) Score 4 = severe (severe/coarse scaling covering almost all or all lesions) Based on this scale, a patient was considered as IGA mod 2011 0/1 responder if the patient achieved a score of 0 or 1 and improved by at least 2 points on the IGA scale compared to baseline.
Time Frame: Week 52, Week 104, Week 156, week 208, week 260
Population: FAS
Measure: Number; unit: Number of participants
Arm/Group | AIN457 150 mg Only | AIN457 300 mg Only
Number analyzed (Participants) | 164 | 416
Number of participants
  Wk 52 | 94 | 311
  Wk 104: number analyzed (Participants) | 104 | 377
  Wk 104 | 63 | 239
  Wk 156: number analyzed (Participants) | 69 | 361
  Wk 156 | 50 | 206
  Wk 208: number analyzed (Participants) | 58 | 323
  Wk 208 | 47 | 183
  Wk 260: number analyzed (Participants) | 51 | 285
  Wk 260 | 39 | 162

9. Secondary Outcome: Percent of Participants With Loss of IGA Mod 2011 0 or 1 Response Over Time for Subjects With IGA Mod 2011 0 or 1 Response at Week 52 - Randomized Withdrawal Period
Description: Summary for loss of IGA mod 2011 0 or 1 response over time for patients with response at Week 52.
  time = 0 refers to Week 52
Time Frame: Week 68
Population: FAS
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | AIN457 150 mg -Randomized Withdrawal Period | AIN457 300 mg -Randomized Withdrawal Period | AIN457 150 mg Placebo - Randomized Withdrawal Period | AIN457 300 mg Placebo - Randomized Withdrawal Period
Number analyzed (Participants) | 297 | 363 | 150 | 180
Percent of participants | 38.1 [29.8 to 47.7] | 33.4 [25.7 to 42.6] | 82.1 [71.2 to 90.8] | 65.5 [53.8 to 77.0]

10. Secondary Outcome: Percent of Participants With PASI 75 Response - Treatment Period for Re-treated After Relapse
Description: PASI 75 response since reinitiating treatment after relapse. time = 0 refers to Week 52
Time Frame: up to week 260
Population: FAS
Measure: Number (95% Confidence Interval); unit: Percent of participants
Groups:
- Placebo - AIN457 150 mg: Patients randomized to placebo at Week 52, treated with AIN457 150mg after they relapsed
- Placebo - AIN457 300 mg: Patients randomized to placebo at Week 52, treated with AIN457 300mg after they relapsed
Arm/Group | Placebo - AIN457 150 mg | Placebo - AIN457 300 mg
Number analyzed (Participants) | 131 | 145
Percent of participants
  0 to <=4 wks | 38.5 [30.7 to 47.4] | 51.0 [43.2 to 59.5]
  >12 to <=16 wks (n=21,13): number analyzed (Participants) | 21 | 13
  >12 to <=16 wks (n=21,13) | 91.2 [85.5 to 95.3] | 95.1 [90.7 to 97.8]
  >80 to <=84 wks (n=2,1): number analyzed (Participants) | 2 | 1
  >80 to <=84 wks (n=2,1) | 96.8 [92.6 to 98.9] | 98.8 [94.8 to 99.9]

11. Secondary Outcome: Percent of Participants With IGA Mod 0 or 1 Response - Treatment Period for Re-treated After Relapse
Description: IGA mod 2011 0 or 1 response since reinitiating treatment after relapse for subjects with IGA 0 or 1 response at week 52 and not have IGA 0 or 1 response at relapse.
  time = 0 refers to Week 52
Time Frame: up to week 260
Population: FAS
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Placebo - AIN457 150 mg | Placebo - AIN457 300 mg
Number analyzed (Participants) | 131 | 145
Percent of participants
  0 to <=4 wks (n=96,123): number analyzed (Participants) | 96 | 123
  0 to <=4 wks (n=96,123) | 12.5 [7.3 to 21.0] | 28.1 [21.0 to 37.0]
  >12 to <=16 wks (n=40,32): number analyzed (Participants) | 40 | 32
  >12 to <=16 wks (n=40,32) | 75.0 [66.0 to 83.1] | 83.5 [76.3 to 89.4]
  >84 to <=88 wks (n=7,4): number analyzed (Participants) | 7 | 4
  >84 to <=88 wks (n=7,4) | 87.9 [80.0 to 93.8] | 90.8 [84.5 to 95.4]

12. Secondary Outcome: Percent pf Participants With Relapse Over Time - Randomized Withdrawal Period
Description: Time 0 = week 52
Time Frame: up to week 156
Population: FAS
Measure: Number (95% Confidence Interval); unit: Percent of participants with relapses
Arm/Group | AIN457 150 mg -Randomized Withdrawal Period | AIN457 300 mg -Randomized Withdrawal Period | AIN457 150 mg Placebo - Randomized Withdrawal Period | AIN457 300 mg Placebo - Randomized Withdrawal Period
Number analyzed (Participants) | 297 | 363 | 150 | 180
Percent of participants with relapses
  0 to <=4 wks (n=286,353,150,180): number analyzed (Participants) | 286 | 353 | 150 | 180
  0 to <=4 wks (n=286,353,150,180) | 0.3 [0.0 to 2.4] | 0.3 [0.0 to 1.9] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
  >12 to <=16 wks (n=297,363,124,160): number analyzed (Participants) | 297 | 363 | 124 | 160
  >12 to <=16 wks (n=297,363,124,160) | 3.1 [1.6 to 5.9] | 2.2 [1.1 to 4.4] | 19.8 [13.9 to 27.7] | 12.1 [8.0 to 18.1]
  >92 to <=96 wks (n=188,292,11,15): number analyzed (Participants) | 188 | 292 | 11 | 15
  >92 to <=96 wks (n=188,292,11,15) | 21.5 [16.9 to 27.0] | 9.4 [6.8 to 13.1] | 88.1 [80.9 to 93.5] | 86.1 [79.6 to 91.4]
  >104 to <=108 wks (n=156,297,8,9): number analyzed (Participants) | 156 | 297 | 8 | 9
  >104 to <=108 wks (n=156,297,8,9) | 21.9 [17.3 to 27.5] | 9.4 [6.8 to 13.1] | 88.1 [80.9 to 93.5] | 86.1 [79.6 to 91.4]

13. Secondary Outcome: Percent of Participants With Relapse After Last Injection
Description: Relapse: when the achieved maximal PASI improvement from baseline of core study was reduced by >50%.
  Time 0 = week 52
Time Frame: up to week 16
Population: FAS
Measure: Number (95% Confidence Interval); unit: Percent of participants with relapse
Arm/Group | AIN457 150 mg Only | AIN457 300 mg Only
Number analyzed (Participants) | 164 | 416
Percent of participants with relapse
  0 to <=4 wks (n=158,415): number analyzed (Participants) | 158 | 415
  0 to <=4 wks (n=158,415) | 7.2 [4.0 to 12.6] | 2.0 [1.0 to 3.9]
  >12 to <=16 wks (n=66,208): number analyzed (Participants) | 66 | 208
  >12 to <=16 wks (n=66,208) | 34.0 [22.6 to 48.9] | 28.4 [21.8 to 36.6]

14. Secondary Outcome: Percent of Participants With Rebound After Last Injection
Description: Rebound: PASI increases to > 125% of baseline (where baseline is the PASI at the randomization of the core study) or presence of new pustular psoriasis, new erythrodermic psoriasis or more inflammatory psoriasis occurring within 8 Weeks of stopping therapy (after the last dose of study treatment received). Rebound like event (RLE) was defined as increase of PASI of > 125% from baseline value or occurrence of new pustular, new erythrodermic or more inflammatory psoriasis any time after stopping therapy (last treatment administered) up to Week 68. Rebound was evaluated for the patients randomized to the placebo groups in the extension study; hence these patients received the last dose of secukinumab during the core studies.
Time Frame: up to week 68
Population: FAS
Measure: Number (95% Confidence Interval); unit: Percent of participants with rebound
Arm/Group | AIN457 150 mg Only | AIN457 300 mg Only
Number analyzed (Participants) | 164 | 416
Percent of participants with rebound
  Rebound (<8 wks after last inj.; n=108,320): number analyzed (Participants) | 108 | 320
  Rebound (<8 wks after last inj.; n=108,320) | 8.3 [4.1 to 15.6] | 6.6 [4.2 to 10.0]
  RLE (< 12 wks after last inj., n=110,326): number analyzed (Participants) | 110 | 326
  RLE (< 12 wks after last inj., n=110,326) | 11.8 [6.7 to 19.7] | 9.5 [6.7 to 13.4]

15. Secondary Outcome: Number of Participants With Dermatology Life Quality Index Response (DLQI 0 or 1) - Randomized Withdrawal Period (Observed Data)
Description: Dermatology Life Quality Index (DLQI) scores range from 0 to 30. Lower absolute scores on DLQI indicate better/improved health-related quality-of life impairment.
Time Frame: Week 52 (baseline), 64, 76, 88, 104, 116, 128, 140, and 156
Population: FAS
Measure: Number; unit: Number of participants
Arm/Group | AIN457 150 mg -Randomized Withdrawal Period | AIN457 300 mg -Randomized Withdrawal Period | AIN457 150 mg Placebo - Randomized Withdrawal Period | AIN457 300 mg Placebo - Randomized Withdrawal Period
Number analyzed (Participants) | 295 | 359 | 150 | 180
Number of participants
  Week 52 (baseline) | 196 | 281 | 109 | 142
  Week 64: number analyzed (Participants) | 290 | 357 | 126 | 162
  Week 64 | 170 | 265 | 59 | 90
  Week 76: number analyzed (Participants) | 284 | 352 | 71 | 104
  Week 76 | 163 | 256 | 26 | 38
  Week 88: number analyzed (Participants) | 281 | 346 | 34 | 62
  Week 88 | 157 | 247 | 18 | 24
  Week 104: number analyzed (Participants) | 262 | 337 | 21 | 35
  Week 104 | 146 | 237 | 10 | 14
  Week 116: number analyzed (Participants) | 252 | 326 | 16 | 24
  Week 116 | 141 | 230 | 6 | 9
  Week 128: number analyzed (Participants) | 251 | 326 | 14 | 19
  Week 128 | 139 | 222 | 4 | 10
  Week 140: number analyzed (Participants) | 241 | 327 | 12 | 18
  Week 140 | 126 | 229 | 4 | 7
  Week 156: number analyzed (Participants) | 240 | 324 | 11 | 15
  Week 156 | 119 | 215 | 5 | 8

16. Secondary Outcome: Number of Participants With Dermatology Life Quality Index Response (DLQI 0 or 1) - Entire Treatment Period
Description: as for outcome 15
Time Frame: Week 52 (baseline), 64, 76, 88, 104, 116, 128, 140, and 156
Population: FAS
Measure: Number; unit: Number of participants
Arm/Group | AIN457 150 mg Only | AIN457 300 mg Only
Number analyzed (Participants) | 164 | 416
Number of participants
  Week 52 (baseline): number analyzed (Participants) | 162 | 412
  Week 52 (baseline) | 95 | 299
  Week 104: number analyzed (Participants) | 113 | 377
  Week 104 | 66 | 254
  week 156: number analyzed (Participants) | 69 | 362
  week 156 | 47 | 225
  Week 208: number analyzed (Participants) | 53 | 328
  Week 208 | 41 | 207
  week 260: number analyzed (Participants) | 52 | 286
  week 260 | 42 | 174

17. Secondary Outcome: EQ-5D Health State Assessment (Observed Value) - Randomized Withdrawal Period
Description: EQ-5D: EuroQOL 5-Dimension Health Status Questionnaire. The EQ-5D© is a generic instrument to assess each patient's health status. It provides a simple descriptive profile and a single index value for health status. The EQ visual analog scale records the respondent's self-rated health on a vertical scale where the endpoints are labeled 'Best imaginable health state' and 'Worst imaginable health state'. This information can be used as a quantitative measure of health outcome as judged by the individual respondents.
Time Frame: Week 52 (baseline), 64, 76, 88, 104, 116, 128, 140, and 156
Population: FAS
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | AIN457 150 mg -Randomized Withdrawal Period | AIN457 300 mg -Randomized Withdrawal Period | AIN457 150 mg Placebo - Randomized Withdrawal Period | AIN457 300 mg Placebo - Randomized Withdrawal Period
Number analyzed (Participants) | 297 | 363 | 150 | 180
Percent change
  Week 64: number analyzed (Participants) | 283 | 348 | 125 | 162
  Week 64 | 0.03 (21.603) | 2.09 (28.358) | -9.58 (20.339) | -5.57 (27.889)
  Week 76: number analyzed (Participants) | 256 | 337 | 72 | 103
  Week 76 | 0.79 (25.605) | 2.76 (29.715) | -13.73 (23.295) | -9.27 (35.302)
  Week 88: number analyzed (Participants) | 241 | 323 | 34 | 60
  Week 88 | 0.07 (21.421) | 2.15 (29.702) | -10.24 (26.026) | -14.67 (27.975)
  Week 104: number analyzed (Participants) | 214 | 310 | 21 | 36
  Week 104 | 2.37 (24.075) | 1.57 (23.941) | -2.81 (27.303) | -9.65 (17.794)
  Week 116: number analyzed (Participants) | 205 | 295 | 16 | 23
  Week 116 | 2.12 (31.724) | 2.06 (24.814) | -4.82 (20.921) | -3.44 (11.846)
  Week 128: number analyzed (Participants) | 201 | 292 | 14 | 19
  Week 128 | 2.06 (33.078) | 3.17 (29.615) | -5.59 (21.756) | -5.97 (13.207)
  Week 140: number analyzed (Participants) | 189 | 288 | 12 | 18
  Week 140 | 1.20 (25.801) | 0.71 (18.151) | -5.90 (27.335) | -8.86 (18.344)
  Week 156: number analyzed (Participants) | 180 | 284 | 11 | 15
  Week 156 | 2.53 (34.259) | 2.23 (22.581) | 3.68 (26.836) | -7.60 (20.683)

18. Secondary Outcome: EQ-5D Health State Assessment (Observed Value) - Entire Study Period
Description: as for outcome 17
Time Frame: week 64, 76, 88, 104, 116, 128, 140, and 156
Population: FAS
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | AIN457 150 mg Only | AIN457 300 mg Only
Number analyzed (Participants) | 164 | 416
Percent change
  Week 64: number analyzed (Participants) | 155 | 404
  Week 64 | -1.33 (22.506) | 1.44 (26.815)
  Week 76: number analyzed (Participants) | 144 | 398
  Week 76 | -1.99 (22.339) | 2.10 (28.493)
  Week 88: number analyzed (Participants) | 130 | 387
  Week 88 | -0.66 (24.558) | 1.45 (28.269)
  Week 104: number analyzed (Participants) | 112 | 376
  Week 104 | -4.15 (27.823) | 0.65 (23.454)
  Week 116: number analyzed (Participants) | 93 | 364
  Week 116 | -1.19 (21.022) | 1.21 (23.681)
  Week 128: number analyzed (Participants) | 84 | 365
  Week 128 | -2.85 (23.584) | 1.93 (27.840)
  Week 140: number analyzed (Participants) | 75 | 367
  Week 140 | 0.09 (20.814) | -0.44 (18.504)
  Week 156: number analyzed (Participants) | 67 | 365
  Week 156 | 2.13 (32.326) | 1.19 (21.548)

19. Secondary Outcome: Clinical Laboratory Evaluation - Hematology Parameters: Incidence Rate for Participants With Clinically CTCAE - Randomized Withdrawal Period
Description: CTCAE: common terminology criteria for adverse events. A subject with multiple variable measurements is counted only once under the worst condition. LLN = lower limit of normal.
  IR=incidence rate per 100 subject years
Time Frame: Week 52-156
Population: Safety set
Measure: Number (95% Confidence Interval); unit: IR
Arm/Group | AIN457 150 mg -Randomized Withdrawal Period | AIN457 300 mg -Randomized Withdrawal Period | AIN457 150 mg Placebo - Randomized Withdrawal Period | AIN457 300 mg Placebo - Randomized Withdrawal Period
Number analyzed (Participants) | 301 | 363 | 150 | 181
IR
  Leukocytes (< LLN - 3.0 x 10E9/L) | 7.0 [4.7 to 10.1] | 4.9 [3.3 to 7.0] | 7.2 [2.6 to 15.6] | 8.6 [4.1 to 15.8]
  Leukocytes (< 3.0 - 2.0 x 10E9/L) | 1.4 [0.5 to 3.0] | 0.8 [0.3 to 1.9] | 0.0 [0.0 to 4.3] | 0.0 [0.0 to 3.1]
  Leukocytes (< 2.0 - 1.0 x 10E9/L) | 0.2 [0.0 to 1.3] | 0.0 [0.0 to 0.6] | 0.0 [0.0 to 4.3] | 0.0 [0.0 to 3.1]
  Leukocytes (< 1.0 x 10E9/L) | 0.0 [0.0 to 0.8] | 0.0 [0.0 to 0.6] | 0.0 [0.0 to 4.3] | 0.0 [0.0 to 3.1]
  Lymphocytes (<LLN-0.8x10e9 /L) | 6.4 [4.2 to 9.4] | 6.1 [4.3 to 8.5] | 4.9 [1.3 to 12.6] | 6.0 [2.4 to 12.4]
  Lymphocytes (<0.8-0.5x10e9 /L) | 3.0 [1.6 to 5.2] | 1.8 [0.9 to 3.2] | 6.3 [2.1 to 14.7] | 3.4 [0.9 to 8.6]
  Lymphocytes (<0.5-0.2 x 10e9 /L) | 0.2 [0.0 to 1.3] | 0.0 [0.0 to 0.6] | 0.0 [0.0 to 4.5] | 0.0 [0.0 to 3.1]
  Lymphocytes (<0.2x10e9 /L) | 0.0 [0.0 to 0.8] | 0.0 [0.0 to 0.6] | 0.0 [0.0 to 4.5] | 0.0 [0.0 to 3.1]
  Neutrophils (<LLN-1.5x10e9 /L) | 5.9 [3.8 to 8.7] | 5.6 [3.8 to 7.8] | 8.7 [3.5 to 18.0] | 11.3 [6.0 to 19.3]
  Neutrophils (<1.5-1.0x10e9 /L) | 1.4 [0.5 to 3.0] | 1.8 [0.9 to 3.2] | 2.4 [0.3 to 8.8] | 0.0 [0.0 to 3.1]
  Neutrophils (<1.0 - 0.5x10e9 /L) | 0.9 [0.3 to 2.4] | 0.5 [0.1 to 1.4] | 0.0 [0.0 to 4.5] | 0.0 [0.0 to 3.1]
  Neutrophils (<0.5x10e9 /L) | 0.0 [0.0 to 0.8] | 0.0 [0.0 to 0.6] | 0.0 [0.0 to 4.5] | 0.0 [0.0 to 3.1]
  Platelets (LLN-75 x10e9 /L) | 3.3 [1.8 to 5.5] | 3.1 [1.9 to 4.9] | 2.4 [0.3 to 8.6] | 5.4 [2.0 to 11.9]
  Platelets (<75-50 x 10e9 /L) | 0.2 [0.0 to 1.3] | 0.2 [0.0 to 0.9] | 0.0 [0.0 to 4.4] | 0.0 [0.0 to 3.2]
  Platelets (<50-25 x 10e9 /L) | 0.0 [0.0 to 0.8] | 0.0 [0.0 to 0.6] | 0.0 [0.0 to 4.4] | 0.0 [0.0 to 3.2]
  Platelets (<25x10e9 /L) | 0.0 [0.0 to 0.8] | 0.2 [0.0 to 0.9] | 0.0 [0.0 to 4.4] | 0.0 [0.0 to 3.2]

20. Secondary Outcome: Clinical Laboratory Evaluation: Number of Participants With Clinically CTCAE - Entire Study Period
Description: CTCAE: common terminology criteria for adverse events. A subject with multiple variable measurements is counted only once under the worst condition. LLN = lower limit of normal.
Time Frame: approximately 4 years
Population: Safety set: The safety set included all patients who took at least one dose of study treatment during the treatment period. Patients were be analyzed according to treatment received.
Measure: Number; unit: Participants
Groups:
- Any AIN457 150 mg: Safety data from patients while on AIN457 150 mg
- Any AIN457 300 mg: Safety data from patients while on AIN457 300 mg
- Any AIN457: safety data from patients while on any dose of AIN457
Arm/Group | Any AIN457 150 mg | Any AIN457 300 mg | Any AIN457
Number analyzed (Participants) | 545 | 890 | 1113
Participants
  Leukocytes (<LLN-3.0x10e9 /L): number analyzed (Participants) | 545 | 832 | 1037
  Leukocytes (<LLN-3.0x10e9 /L) | 55 | 59 | 114
  Leukocytes (<3.0-2.0 x 10e9 /L): number analyzed (Participants) | 545 | 866 | 1080
  Leukocytes (<3.0-2.0 x 10e9 /L) | 10 | 7 | 17
  Leukocytes (<2.0-1.0x10e9 /L): number analyzed (Participants) | 545 | 870 | 1085
  Leukocytes (<2.0-1.0x10e9 /L) | 1 | 0 | 1
  Leukocytes (<1.0x10e9 /L): number analyzed (Participants) | 545 | 870 | 1085
  Leukocytes (<1.0x10e9 /L) | 0 | 0 | 0
  Lymphocytes (<LLN-0.8x10e9 /L): number analyzed (Participants) | 545 | 840 | 1041
  Lymphocytes (<LLN-0.8x10e9 /L) | 47 | 61 | 108
  Lymphocytes (<0.8-0.5x10e9 /L): number analyzed (Participants) | 545 | 861 | 1071
  Lymphocytes (<0.8-0.5x10e9 /L) | 18 | 28 | 46
  Lymphocytes (<0.5-0.2 x 10e9 /L, n=545,864,1075): number analyzed (Participants) | 545 | 864 | 1075
  Lymphocytes (<0.5-0.2 x 10e9 /L, n=545,864,1075) | 1 | 1 | 2
  Lymphocytes (<0.2x10e9 /L, n=545,864,1075): number analyzed (Participants) | 545 | 864 | 1075
  Lymphocytes (<0.2x10e9 /L, n=545,864,1075) | 0 | 0 | 0
  Neutrophils (<LLN-1.5x10e9 /L): number analyzed (Participants) | 545 | 831 | 1037
  Neutrophils (<LLN-1.5x10e9 /L) | 54 | 69 | 123
  Neutrophils (<1.5-1.0x10e9 /L): number analyzed (Participants) | 545 | 861 | 1071
  Neutrophils (<1.5-1.0x10e9 /L) | 12 | 20 | 32
  Neutrophils (<1.0 - 0.5x10e9 /L,): number analyzed (Participants) | 545 | 863 | 1074
  Neutrophils (<1.0 - 0.5x10e9 /L,) | 7 | 4 | 11
  Neutrophils (<0.5x10e9 /L): number analyzed (Participants) | 545 | 864 | 1075
  Neutrophils (<0.5x10e9 /L) | 0 | 0 | 0
  Platelets (LLN-75x10e9 /L): number analyzed (Participants) | 545 | 836 | 1042
  Platelets (LLN-75x10e9 /L) | 24 | 39 | 63
  Platelets (<75-50x10e9 /L,): number analyzed (Participants) | 545 | 862 | 1074
  Platelets (<75-50x10e9 /L,) | 2 | 2 | 4
  Platelets (<50-25 x 10e9 /L): number analyzed (Participants) | 545 | 862 | 1074
  Platelets (<50-25 x 10e9 /L) | 0 | 0 | 0
  Platelets (<25x10e9 /L): number analyzed (Participants) | 545 | 862 | 1074
  Platelets (<25x10e9 /L) | 0 | 1 | 1

21. Secondary Outcome: Electrocardiogram: Incidence of Participants With ECG Test Results - Randomized Withdrawal Period
Description: QTcB: QT interval corrected using Bazett's formula QTcF: QT interval corrected using Fridericia's formula A patient with multiple variable measurements is counted only once under the worst condition.
  IR=incidence rate per 100 subject years.
Time Frame: Week 52 - 156
Population: Safety set
Measure: Number (95% Confidence Interval); unit: IR
Arm/Group | AIN457 150 mg -Randomized Withdrawal Period | AIN457 300 mg -Randomized Withdrawal Period | AIN457 150 mg Placebo - Randomized Withdrawal Period | AIN457 300 mg Placebo - Randomized Withdrawal Period
Number analyzed (Participants) | 301 | 363 | 150 | 181
IR
  QTcB>450 msec | 10.5 [7.5 to 14.3] | 9.4 [7.0 to 12.4] | 11.3 [4.9 to 22.3] | 14.1 [7.5 to 24.0]
  QTcB>480 msec | 0.7 [0.1 to 2.0] | 1.1 [0.5 to 2.3] | 0.0 [0.0 to 4.7] | 0.0 [0.0 to 3.3]
  QTcB>500 msec | 0.2 [0.0 to 1.3] | 0.2 [0.0 to 0.9] | 0.0 [0.0 to 4.7] | 0.0 [0.0 to 3.3]
  QTcB change from baseline>30 ms | 15.6 [11.9 to 20.1] | 14.3 [11.4 to 17.9] | 21.6 [12.3 to 35.0] | 15.7 [9.0 to 25.5]
  QTcB change from baseline>60 ms | 0.7 [0.1 to 2.0] | 0.8 [0.3 to 1.9] | 0.0 [0.0 to 4.7] | 0.0 [0.0 to 3.3]
  QTcF>450 msec | 3.6 [2.0 to 6.0] | 3.0 [1.8 to 4.7] | 2.6 [0.3 to 9.5] | 4.7 [1.5 to 10.9]
  QTcF>480 msec | 0.5 [0.1 to 1.7] | 0.2 [0.0 to 0.9] | 0.0 [0.0 to 4.7] | 0.9 [0.0 to 5.0]
  QTcF>500 msec | 0.0 [0.0 to 0.8] | 0.0 [0.0 to 0.6] | 0.0 [0.0 to 4.7] | 0.0 [0.0 to 3.3]
  QTcF change from baseline>30 ms | 6.9 [4.6 to 9.9] | 6.8 [4.8 to 9.2] | 7.9 [2.9 to 17.2] | 9.5 [4.6 to 17.5]
  QTcF change from baseline>60 ms | 0.2 [0.0 to 1.3] | 0.2 [0.0 to 0.9] | 0.0 [0.0 to 4.7] | 0.0 [0.0 to 3.3]
  PR>250 msec | 0.2 [0.0 to 1.3] | 0.0 [0.0 to 0.6] | 0.0 [0.0 to 4.9] | 0.0 [0.0 to 3.3]

22. Secondary Outcome: Electrocardiogram: Number of Participants With ECG Test Results - Entire Treatment Period
Description: QTcB: QT interval corrected using Bazett's formula QTcF: QT interval corrected using Fridericia's formula A patient with multiple variable measurements is counted only once under the worst condition.
Time Frame: Approximately 4 years
Population: Safety set
Measure: Number; unit: Participants
Arm/Group | Any AIN457 150 mg | Any AIN457 300 mg | Any AIN457
Number analyzed (Participants) | 545 | 890 | 1113
Participants
  QTcB>500 msec: number analyzed (Participants) | 545 | 851 | 1060
  QTcB>500 msec | 1 | 2 | 3
  QTcB>480 msec: number analyzed (Participants) | 545 | 848 | 1056
  QTcB>480 msec | 8 | 23 | 30
  QTcB>450 msec: number analyzed (Participants) | 545 | 804 | 1004
  QTcB>450 msec | 86 | 159 | 218
  QTcB changes from baseline>30 ms: number analyzed (Participants) | 545 | 851 | 1060
  QTcB changes from baseline>30 ms | 124 | 223 | 316
  QTcB changes from baseline>60 ms: number analyzed (Participants) | 545 | 851 | 1060
  QTcB changes from baseline>60 ms | 7 | 19 | 25
  QTcF>500 msec: number analyzed (Participants) | 545 | 851 | 1060
  QTcF>500 msec | 0 | 1 | 1
  QTcF>480 msec: number analyzed (Participants) | 545 | 851 | 1059
  QTcF>480 msec | 3 | 6 | 8
  QTcF>450 msec (n=545,838,1043): number analyzed (Participants) | 545 | 838 | 1043
  QTcF>450 msec (n=545,838,1043) | 35 | 67 | 93
  QTcF changes from baseline>30 ms: number analyzed (Participants) | 545 | 851 | 1060
  QTcF changes from baseline>30 ms | 69 | 127 | 184
  QTcF changes from baseline>60 ms: number analyzed (Participants) | 545 | 851 | 1060
  QTcF changes from baseline>60 ms | 1 | 3 | 4
  PR>250 msec: number analyzed (Participants) | 545 | 845 | 1051
  PR>250 msec | 4 | 5 | 8

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All AEs reported in this record are from date of First Patient First Treatment until Last Patient Last Visit) up to approximately 5 years.
Description: Consistent with EudraCT disclosure specifications, Novartis has reported under the Serious adverse events fields "number of deaths resulting from adverse events" all those deaths, resulting from serious adverse events that are deemed to be causally related to treatment by the investigator.
Groups:
- Any AIN457 Dose: safety data from patients while on any dose of AIN457
- AIN457 150 mg - Placebo; AIN457 300 mg - Placebo: safety data from patients of corresponding randomized withdrawal group while on placebo
Arm/Group | Any AIN457 150 mg | Any AIN457 300 mg | Any AIN457 Dose | AIN457 150 mg - Placebo | AIN457 300 mg - Placebo
All-Cause Mortality (participants affected / at risk) | 0/545 | 2/890 | 2/1113 | 0/150 | 0/181
Serious Adverse Events (participants affected / at risk) | 61/545 | 143/890 | 198/1113 | 4/150 | 13/181
Other Adverse Events (participants affected / at risk) | 386/545 | 679/890 | 889/1113 | 75/150 | 86/181
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Any AIN457 150 mg (N=545) | Any AIN457 300 mg (N=890) | Any AIN457 Dose (N=1113) | AIN457 150 mg - Placebo (N=150) | AIN457 300 mg - Placebo (N=181)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 0
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 4 | 4 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 4 | 4 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 1 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 9 | 10 | 0 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 1 | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 1 | 3 | 4 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 2 | 3 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 1 | 0 | 0
Stress cardiomyopathy (Cardiac disorders) | 0 | 1 | 1 | 0 | 0
Tachycardia paroxysmal (Cardiac disorders) | 1 | 0 | 1 | 0 | 0
Ventricular fibrillation (Cardiac disorders) | 1 | 0 | 1 | 0 | 0
Malformation venous (Congenital, familial and genetic disorders) | 0 | 1 | 1 | 0 | 0
Hyperandrogenism (Endocrine disorders) | 1 | 0 | 1 | 0 | 0
Thyroid mass (Endocrine disorders) | 0 | 1 | 1 | 0 | 0
Cataract (Eye disorders) | 1 | 0 | 1 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 1 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1
Diverticulum (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 2 | 2 | 0 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Functional gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 1 | 2 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Ileus paralytic (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 2 | 2 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Intestinal polyp (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Large intestinal stenosis (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 2 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Umbilical hernia, obstructive (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 1 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 1
Face oedema (General disorders) | 0 | 1 | 1 | 0 | 0
Impaired healing (General disorders) | 0 | 1 | 1 | 0 | 0
Medical device site granuloma (General disorders) | 0 | 1 | 1 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 1 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 2 | 2 | 0 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 1 | 1 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 1 | 1 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 1 | 0 | 0
Cholangitis acute (Hepatobiliary disorders) | 0 | 1 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 2 | 2 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 2 | 2 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 1 | 3 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 1 | 0 | 1 | 0 | 0
Hepatitis acute (Hepatobiliary disorders) | 0 | 1 | 1 | 0 | 0
Hepatitis toxic (Hepatobiliary disorders) | 0 | 1 | 1 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 1 | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 1 | 0 | 0
Sarcoidosis (Immune system disorders) | 0 | 0 | 0 | 0 | 1
Abscess limb (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Abscess neck (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Acute sinusitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 2 | 2 | 4 | 0 | 2
Appendicitis perforated (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 2 | 2 | 1 | 1
Cholecystitis infective (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Chronic sinusitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Chronic tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Device related infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 3 | 1 | 4 | 0 | 1
Enterococcal bacteraemia (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Epididymitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 1 | 0 | 1
Escherichia infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Gallbladder empyema (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Graft infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Hepatitis A (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Implant site infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Localised infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Oophoritis (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Otitis media (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Periorbital cellulitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Peritonitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Peritonsillar abscess (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Pharyngeal abscess (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 4 | 5 | 0 | 0
Pneumonia influenzal (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Post procedural infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 4 | 4 | 0 | 0
Septic shock (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 1 | 2 | 0 | 0
Streptococcal infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Tick-borne viral encephalitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 2 | 2 | 4 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 2 | 0 | 0
Viral pericarditis (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Wound infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Accident (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 1 | 3 | 0 | 1
Cardiac procedure complication (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 3 | 3 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0
Kidney rupture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0
Ligament injury (Injury, poisoning and procedural complications) | 0 | 2 | 2 | 0 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 2 | 3 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 2 | 2 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 3 | 3 | 0 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 2 | 2 | 0 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 2 | 2 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0
Procedural hypertension (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 2 | 2 | 0 | 1
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0
Tendon injury (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 3 | 3 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 2 | 3 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1 | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 1
Joint instability (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3 | 0 | 0
Osteitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 4 | 5 | 0 | 0
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0
Anal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 3 | 0 | 0
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Complex regional pain syndrome (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Cranial nerve paralysis (Nervous system disorders) | 1 | 0 | 1 | 0 | 0
Diabetic neuropathy (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 0 | 0
Drooling (Nervous system disorders) | 1 | 0 | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Intracranial aneurysm (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Lumbar radiculopathy (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Parkinson's disease (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 1 | 0 | 1
Tremor (Nervous system disorders) | 1 | 0 | 1 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 1 | 0 | 0
Abortion spontaneous complete (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 1 | 0 | 0
Device dislocation (Product Issues) | 1 | 0 | 1 | 0 | 0
Device loosening (Product Issues) | 0 | 1 | 1 | 0 | 0
Alcoholism (Psychiatric disorders) | 1 | 1 | 2 | 0 | 0
Aversion (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0
Completed suicide (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0
Depression (Psychiatric disorders) | 3 | 2 | 5 | 0 | 0
Hypomania (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0
Schizophrenia (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0
Substance abuse (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 2 | 2 | 0 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 0
Nephrotic syndrome (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 0
Urethral stenosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 1 | 1 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 1 | 0 | 0
Vaginal cyst (Reproductive system and breast disorders) | 0 | 1 | 1 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3 | 0 | 0
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0
Sinus polyp (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 2 | 3 | 5 | 0 | 0
Circulatory collapse (Vascular disorders) | 0 | 1 | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 2 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 3 | 3 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 1 | 0 | 0
Varicose vein (Vascular disorders) | 0 | 1 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Any AIN457 150 mg (N=545) | Any AIN457 300 mg (N=890) | Any AIN457 Dose (N=1113) | AIN457 150 mg - Placebo (N=150) | AIN457 300 mg - Placebo (N=181)
Abdominal pain upper (Gastrointestinal disorders) | 11 | 15 | 25 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 29 | 53 | 81 | 3 | 5
Gastritis (Gastrointestinal disorders) | 11 | 21 | 31 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 12 | 25 | 37 | 1 | 0
Nausea (Gastrointestinal disorders) | 9 | 15 | 24 | 0 | 0
Toothache (Gastrointestinal disorders) | 10 | 33 | 43 | 0 | 2
Influenza like illness (General disorders) | 24 | 45 | 65 | 2 | 2
Pyrexia (General disorders) | 7 | 24 | 31 | 0 | 2
Seasonal allergy (Immune system disorders) | 8 | 19 | 27 | 2 | 1
Bronchitis (Infections and infestations) | 31 | 63 | 92 | 3 | 3
Conjunctivitis (Infections and infestations) | 10 | 30 | 38 | 1 | 1
Cystitis (Infections and infestations) | 10 | 23 | 31 | 0 | 1
Folliculitis (Infections and infestations) | 13 | 18 | 31 | 1 | 2
Gastroenteritis (Infections and infestations) | 24 | 35 | 59 | 3 | 2
Herpes zoster (Infections and infestations) | 3 | 25 | 27 | 2 | 0
Influenza (Infections and infestations) | 24 | 54 | 78 | 4 | 6
Nasopharyngitis (Infections and infestations) | 145 | 271 | 375 | 17 | 21
Oral candidiasis (Infections and infestations) | 7 | 22 | 29 | 1 | 0
Oral herpes (Infections and infestations) | 12 | 25 | 36 | 2 | 2
Pharyngitis (Infections and infestations) | 18 | 38 | 55 | 1 | 3
Rhinitis (Infections and infestations) | 11 | 30 | 38 | 0 | 1
Sinusitis (Infections and infestations) | 18 | 51 | 64 | 4 | 3
Tinea pedis (Infections and infestations) | 9 | 29 | 38 | 0 | 2
Tonsillitis (Infections and infestations) | 19 | 31 | 49 | 6 | 3
Tooth infection (Infections and infestations) | 10 | 18 | 28 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 52 | 119 | 153 | 8 | 12
Urinary tract infection (Infections and infestations) | 15 | 33 | 46 | 3 | 2
Viral upper respiratory tract infection (Infections and infestations) | 11 | 21 | 31 | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 9 | 22 | 31 | 1 | 2
Laceration (Injury, poisoning and procedural complications) | 9 | 16 | 25 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 13 | 21 | 34 | 1 | 2
Muscle strain (Injury, poisoning and procedural complications) | 9 | 17 | 25 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 8 | 21 | 29 | 1 | 0
Alanine aminotransferase increased (Investigations) | 13 | 8 | 21 | 1 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 3 | 18 | 20 | 1 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 11 | 9 | 20 | 2 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 11 | 18 | 29 | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 47 | 80 | 124 | 8 | 13
Back pain (Musculoskeletal and connective tissue disorders) | 40 | 76 | 114 | 4 | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 14 | 19 | 33 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 10 | 22 | 32 | 3 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 20 | 29 | 49 | 2 | 2
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 11 | 38 | 47 | 8 | 6
Tendonitis (Musculoskeletal and connective tissue disorders) | 5 | 23 | 28 | 1 | 1
Headache (Nervous system disorders) | 36 | 87 | 116 | 4 | 2
Anxiety (Psychiatric disorders) | 8 | 20 | 28 | 1 | 1
Depression (Psychiatric disorders) | 14 | 10 | 24 | 2 | 2
Insomnia (Psychiatric disorders) | 11 | 20 | 30 | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 27 | 43 | 66 | 1 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 23 | 42 | 65 | 3 | 3
Dermatitis contact (Skin and subcutaneous tissue disorders) | 5 | 19 | 23 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 8 | 34 | 41 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 11 | 24 | 34 | 2 | 3
Psoriasis (Skin and subcutaneous tissue disorders) | 14 | 39 | 51 | 1 | 3
Hypertension (Vascular disorders) | 42 | 83 | 119 | 5 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2015-04-29): https://cdn.clinicaltrials.gov/large-docs/95/NCT01544595/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-02): https://cdn.clinicaltrials.gov/large-docs/95/NCT01544595/SAP_001.pdf